CLINICAL TRIAL: NCT00498446
Title: Imaging of Atrial Septal Defects by Velocity Encoded Cardiovascular Magnetic Resonance
Brief Title: Magnetic Resonance Imaging of Atrial Septal Defects
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Other Study IDs: 3938
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2007-07

CONDITIONS: Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
An atrial septal defect (ASD) is a hole in the heart that can lead to heart failure. Depending on the size and severity of the ASD, They can be treated during a heart catheterization with a special device that can permanently seal the ASD, but knowing the exact size and severity of the ASD is crucial. Newer MRI techniques may provide a better way at diagnosing the size and severity of an ASD. We compared MRI to other standard clinical ways for evaluating an ASD.

DETAILED DESCRIPTION:
Background: Atrial septal defect (ASD) flow can be measured indirectly by velocity-encoded cardiovascular magnetic resonance (veCMR) of the pulmonary artery and aorta (Qp/Qs). Imaging the secundum ASD en face could potentially enable direct flow measurement and, additionally, provide valuable information regarding ASD size, shape, location, and proximity to other structures.

Methods: Patients referred for possible transcatheter ASD closure underwent a comprehensive standard evaluation including transesophageal and/or intracardiac echocardiography (ICE), and invasive oximetry. CMR was performed in parallel and included direct en face veCMR after an optimal double-oblique imaging plane was determined accounting for ASD flow direction and cardiac-cycle interatrial septal motion.

We hypothesized that En face veCMR using an optimized imaging plane can accurately determine ASD flow, size, and morphology, and that it would provide information incremental to comprehensive standard evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Suspected Atrial Septal Defect (ASD) undergoing evaluation for possible transcatheter closure

Exclusion Criteria:

* Contraindications to magnetic resonance imaging
* known sinus venosus or primum defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-07; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J Kim, MD, Principal Investigator — Duke Cardiovascular Magnetic Resonance Center
Locations (1):
- Duke Cardiovascular Magnetic Resonance Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Thomson LE, Crowley AL, Heitner JF, Cawley PJ, Weinsaft JW, Kim HW, Parker M, Judd RM, Harrison JK, Kim RJ. Direct en face imaging of secundum atrial septal defects by velocity-encoded cardiovascular magnetic resonance in patients evaluated for possible transcatheter closure. Circ Cardiovasc Imaging. 2008 Jul;1(1):31-40. doi: 10.1161/CIRCIMAGING.108.769786. PMID 19808512